CLINICAL TRIAL: NCT06984354
Title: NOTUS Trial: A Randomised Controlled Trial of Two Digitally Delivered Treatment Options for Chronic Back Pain
Brief Title: Digitally Delivered Treatments to Reduce Chronic Low Back Pain
Acronym: NOTUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroscience Research Australia (Other)
Responsible Party: Principal Investigator, James McAuley, Principal Investigator, Neuroscience Research Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iRECS4383
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain; Chronic Pain (Back / Neck); General Practice (GP), Primary Care Settings; Digital Health; Hypnosis, Chronic Pain Management; Patient Education
Keywords: Back Pain; Digital Health; Hypnosis; Pain Education; Chronic Pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Back Pain

STUDY DESIGN:
Masking Description: The statistician will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain education and clinical hypnosis delivered via a mobile app (Experimental): Pain education and clinical hypnosis for self-managing back pain, delivered via a mobile app.
  Interventions: Behavioral: Pain education and clinical hypnosis delivered via a mobile app
- Guideline-informed factsheet (Active Comparator): A guideline-informed factsheet for back pain, delivered via a webpage.
  Interventions: Behavioral: Guideline-informed factsheet

INTERVENTIONS:
Behavioral: Pain education and clinical hypnosis delivered via a mobile app — Pain education and clinical hypnosis will be delivered via a mobile app. The 8-week intervention includes daily sessions on pain education and clinical hypnosis for managing back pain (5 minutes of education, 15 minutes of listening to hypnotherapy audio and engaging in physical/social activities for 5 minutes). The first six weeks will be semi-standardised, with participants following a set program with the option to repeat sessions. The last two weeks will be flexible, allowing participants to choose a specific program or self-paced continuation of the intervention. Adherence will be monitored by tracking the number of days participants complete sessions, as recorded by the mobile app.
  Arms: Pain education and clinical hypnosis delivered via a mobile app
Behavioral: Guideline-informed factsheet — A single guideline-informed factsheet for back pain delivered via a webpage. Participants will be informed that the factsheet intends to provide reassurance for their back pain and encourage reflections on treatments and self-management options.
  Arms: Guideline-informed factsheet

SUMMARY:
This study aims to evaluate the effectiveness of pain education and clinical hypnosis delivered via a mobile app compared to a guideline-informed factsheet for reducing pain and disability in people experiencing chronic low back pain attending general practice.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing non-specific chronic low back pain (LBP), defined as pain between the 12th rib and the buttock crease.
* LBP with or without leg pain (in case of leg pain, LBP is worse than leg pain).
* Currently consulting with a general practitioner for their non-specific chronic LBP across Australia.
* Mean pain intensity score on the Numeric Rating Scale ≥ 3/10 in the past week.
* A score of at least moderate on question 8 of the physical functioning component of the SF-36 questionnaire.
* Access to a mobile device with minimal requirements to download the study app (300MB).
* An internet connection to access the mobile app functionalities.
* Able to understand English via reading and audio materials.

Exclusion Criteria:

* Known or suspected specific spinal (e.g., radiculopathy, fracture) or specific non-spinal non- (e.g., tumour, infection) pathology.
* Less than six months post-spinal surgery.
* Scheduled for major surgery during the program or the follow-up period.
* Known or suspected serious psychiatric condition not being treated by a health professional that would impact adherence to the trial activities.
* Known or suspected sight or hearing problems that would limit access to the intervention components (reading and listening using headphones).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-05-26 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Week 8 post-randomisation
  Average pain intensity over the past 7 days measured using the Numeric Rating Scale, 0 (no pain) to 10 (worst pain imaginable)
Disability | Week 8 post-randomisation
  Disability will be measured using the Roland-Morris Disability Questionnaire scale, ranging from 0 to 24, with higher scores representing higher levels of disability.

SECONDARY OUTCOMES:
Pain intensity | Weeks 12, 26 and 52 post-randomisation
  Average pain intensity over the past 7 days will be measured using the Numeric Rating Scale, 0 (no pain) to 10 (worst pain imaginable).
Disability | Weeks 12, 26 and 52 post-randomisation
  Disability will be measured using the Roland Morris Disability Questionnaire, 0 to 24, with higher scores representing higher levels of disability.
Worst pain intensity | Weeks 8, 12, 26 and 52 post-randomisation
  Worst pain intensity over the past 7 days will be measured using the Numeric Rating Scale, 0 (no pain) to 10 (worst pain imaginable).
Adverse events | Week 8 post-randomisation
  Adverse events will be assessed using self-reported information during the trial.
Health-related quality of life | Weeks 8, 12, 26 and 52 post-randomisation
  Health-related quality of life will be measured using the EuroQol 5-Dimensions 5-Level (EQ-5D-5L) questionnaire, which includes an index score ranging from 0 to 1 and a health visual analogue scale (VAS) ranging from 0 to 100, with higher scores indicating a better health state.
Global impression of change | Weeks 8, 12, 26 and 52 post-randomisation
  Global impression of change measured by the Global Perceived Effect Scale using the following questions: 'With respect to your low back pain, how would you describe yourself now compared to when you started the treatment program?' (range, -5 to 5; lower scores indicate worse outcomes).
Anxiety symptoms | Weeks 8, 12, 26 and 52 post-randomisation
  Anxiety symptoms will be measured by the anxiety sub-scale from the Depression, Anxiety, Stress Scale (DASS-21), scores ranging from 0 to 42, with higher scores indicating worse symptoms.
Depression symptoms | Weeks 8, 12, 26 and 52 post-randomisation
  Depression symptoms will be measured by the depression sub-scale from the Depression, Anxiety, Stress Scale (DASS-21), scores ranging from 0 to 42, with higher scores indicating worse symptoms.

OTHER OUTCOMES:
Cost-utility analysis | From randomisation to week 52 post-randomisation
  The cost-utility of the intervention will be evaluated by calculating quality-adjusted life years using the EuroQOL EQ-5D-5L measure. The total cost of delivering the intervention within the trial will be calculated, along with total healthcare consumption external to the trial, using data from the Medicare and Pharmaceutical Benefits Scheme databases and self-reports.

CONTACTS AND LOCATIONS:
Overall Officials: James H McAuley, PhD, Principal Investigator — Neuroscience Research Australia
Locations (1):
- Neuroscience Research Australia, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to interested researchers only upon reasonable request and once the proposed research project has received separate ethics approval from a Human Research Ethics Committee.
  Request to the data custodian, the Principal Investigator (j.mcauley@neura.edu.au).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available after the publication of the study reports. There is no end date for the availability of study data.
Access Criteria: Protocol and ethics must be provided.